CLINICAL TRIAL: NCT01177085
Title: Substituting Mushrooms for Meat: A Controlled Clinical Trial to Control Body Weight
Brief Title: Substituting Mushrooms for Meat to Control Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mush2
Record Dates: First submitted 2008-11-05; First posted 2010-08-06 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Obesity
Keywords: obesity; weight; weight-loss; mushroom; oxidative; stress; immune; function; inflammation
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mushroom (Experimental): Mushroom enriched weight loss diet. Participants will be given a personalized diet plan, at a calorie level sufficiently restricted to result in a 20 lb weight loss over a period of 6 months, followed by a weight maintenance diet for a further 6 months.
  Interventions: Behavioral: Weight-loss and weight-maintenance diets
- No mushroom diet (Active Comparator): Participants will be given a personalized diet plan, without use of mushrooms as part of the diet, at a calorie level sufficiently restricted to result in a 20 lb weight loss over a period of 6 months, followed by a weight maintenance diet for a further 6 months.
  Interventions: Behavioral: Weight-loss and weight-maintenance diets

INTERVENTIONS:
Behavioral: Weight-loss and weight-maintenance diets — Participants will be given a personalized diet plan, with or without use of mushrooms as part of the diet, at a calorie level sufficiently restricted to result in a 20 lb weight loss over a period of 6 months, followed by a weight maintenance diet for a further 6 months.

SUMMARY:
This is a one-year clinical trial to assess weight-loss, weight-maintenance, and biochemical parameters following a weight-control diet using either standard food guide pyramid alone, or standard food guide pyramid with substitution of mushrooms for meat.

DETAILED DESCRIPTION:
This intervention study has a primary aim to assess omnivorous adult males and females' ability to control their weight over a period of 1 year. The control group will be required to use 90% lean ground beef a few times per week for one year while maintaining their personalized diet plans. The experimental group will have to follow their personalized diets as well, but will be required to substitute mushrooms for meat at least three times per week. Biochemical measures will also be assessed in response to the diet and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, >=18 years old
* Omnivorous
* BMI 25-40
* Seeking weight-loss

Exclusion Criteria:

* <18 years old
* Vegetarians
* Dislike mushroom
* Chronic disease
* HIV+
* Rheumatoid arthritis
* Pregnant or nursing child
* Must not self-report allergies to mushrooms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Weight-control efficacy | 1 year
Weight-loss efficacy | 6 months

SECONDARY OUTCOMES:
Effect of mushroom-substituted meals on biomarkers for oxidative stress, immune function and inflammation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cheskin LJ, Davis LM, Lipsky LM, Mitola AH, Lycan T, Mitchell V, Mickle B, Adkins E. Lack of energy compensation over 4 days when white button mushrooms are substituted for beef. Appetite. 2008 Jul;51(1):50-7. doi: 10.1016/j.appet.2007.11.007. Epub 2007 Dec 3. PMID 18221822